CLINICAL TRIAL: NCT01324817
Title: Substantial Equivalence Study for Kai Medical Non-Contact Respiratory Rate Monitors for Use With Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kai Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: KAI-00006
Record Dates: First submitted 2011-03-26; First posted 2011-03-29 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Respiration
Keywords: Non-Contact; Radar; Doppler; Respiratory; Respiration; Breathing; Rate; Frequency; Respiratory Mechanics; Respiratory Rate Measurement; Apnea; Sleep Apnea
MeSH Terms: conditions — Respiratory Aspiration; Apnea; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hopitalized: Patients admitted to the hospital
  Interventions: Device: Kai Spot (v 2.1); Device: Kai Continuous (v 1.0)

INTERVENTIONS:
Device: Kai Spot (v 2.1) — The Kai Spot (v 2.1) provides a measurement of respiratory rate at a single point in time for neonates, pediatrics, and adults.
  Other Names: Kai Spot
Device: Kai Continuous (v 1.0) — The Kai Continuous (v 1.0) provides a continuous monitor, measurement, and display of the respiratory rate, respiratory patterns, depth of breath, history/events and respiratory activity of a subject for neonates, pediatrics, and adults.
  Other Names: Kai Continuous

SUMMARY:
The purpose of this study is to test the accuracy of two devices (the Kai Spot (v 2.1) and the Kai Continuous (v 1.0) that can measure breathing patters (how fast you breath) without wires and without touching the body.

DETAILED DESCRIPTION:
The purpose of this study is to test two remote, Doppler radar-based sensors to measure and monitor respiratory rate. Specifically, in clinically stable neonatal patients the study aims to:

1. Obtain respiratory effort data of neonatal patients with remote Doppler radar systems modified from a system cleared by the FDA for adult use.
2. Determine if remote Doppler radar systems can accurately detect the respiratory rate of neonatal patients, compared with standard measurement systems.
3. Determine if unattended Doppler radar systems, operating for 4 hours, can accurately detect the respiratory rate of neonatal patients.

ELIGIBILITY:
* Inclusion Criteria:

  1. Clinically stable
* Exclusion Criteria:

  1. Clinically unstable
* Hypotensive requiring pressors
* Intubated

  2. Scheduled or planned (e.g., CT scan, central line placement) procedure during the study period.

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates hospitalized at the Kapiolani Medical Center for Women and Children located in Honolulu, HI
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Venkataraman Balaraman, MD, Principal Investigator — Kapiolani Medical Center For Women & Children
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States